CLINICAL TRIAL: NCT05045976
Title: Efficacy of an Interactive Web-based Self-management Support Intervention on Health Outcomes in Patients With Colorectal Cancer: A Mixed-methods Study
Brief Title: Efficacy of Web-based Self-management Support Intervention on Health Outcomes in Patients With Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Mackay Memorial Hospital (Other); Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, Director, School of Nursing, National Taipei University of Nursing and Health Sciences, Taipei, Taiwan, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NTUNHS-107EH12-37
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; web-based interactive self-management support; health-related quality of life; self-efficacy; emotion distress; supportive care needs; symptom distress; healthy life styles
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study participants will be randomly assigned 1:1 to the intervention or the control group by the stratified permuted block randomization and block 4, 6, 8 will be used. The randomization will be stratified by cancer stage (stage I-IIA; stage IIB-III). The Sealed Envelope software (Sealed Envelope Ltd., 2016) will be used to generate the random sequences and sealed envelopes will be used to conceal the assignment of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive the web-based interactive self-management support intervention.
  Interventions: Other: Web-based interactive self-management support program
- Control group (No Intervention): The control group will receive usual care and regular patients education.

INTERVENTIONS:
Other: Web-based interactive self-management support program — The intervention group will receive a 60-90 minute introduction to the web-based interactive self-management support program. They will be instructed to do the weekly online self-assessment on symptoms, emotion, and health behaviors and how to use the web-based program to manage their health by applying self-manage skills and behavior change techniques. The contents of the interactive colorectal cancer self-management website include the following five main components: Health Support Station, Knowledge Supply Station, Sharing Stories, My Dear Friend, and Asking a Nurse.
  Arms: Experimental group

SUMMARY:
The study aims to test the efficacy of a web-based interactive self-management support intervention on the primary outcome, quality of life, secondary outcomes, symptom distress, emotional distress, physical activity, and the mediation effects of self-efficacy, and supportive care needs in colorectal cancer patients.

DETAILED DESCRIPTION:
Colorectal cancer is the most commonly diagnosed cancer in Taiwan. With proper treatments, most patients can be long-term survivors. However, patients often suffered long-term consequences of the disease and its treatment side effects. In addition, unhealthy lifestyles will further impact on patient's prognosis and quality of life. Face-to-face or web-based self-management support interventions can help colorectal cancer patients to achieve a healthy lifestyle and better adjustment. However, they are costly and may not be assessable for a certain population. Therefore, it is necessary to develop the most cost-effective interventions for patients with colorectal cancer.

Aim: The study aims is to test the efficacy of a web-based interactive self-management support intervention on the primary outcome, quality of life, and secondary outcomes, symptom distress, emotional distress, physical activity, nutrition intake, and the mediation effects of self-efficacy, social support, and supportive care needs in colorectal cancer patients.

Design: A multi-center randomized six-month follow-up parallel-group superiority design will be used to test the intervention efficacy. A convenient sample of 160 post-operative colorectal cancer patients (stage I-III) will be recruited and randomized to the control or intervention group. Outcome variables will be assessed on the baseline, 2nd, 4th, and 6th month in both groups.

Instruments: The study instruments include Cancer Behavior Inventory-Brief Version, 34-item Supportive Care Needs Survey, M.D. Anderson Symptom Inventory, The Center for Epidemiologic Studies Depression Scale, International Physical Activity Questionnaire, and FACT-C.

Data analysis: Descriptive analysis will be used to describe patients' demographics, disease variables, and outcome variables. The Chi-square, t-test, and Linear Mixed Model will be used to test the efficacy of the study interventions.

Significance: The study results will provide evidence for the efficacy of the web-based interactive self-management support intervention for enhancing a healthy lifestyle and quality of life in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer (ICD-10 code: C18-C20, C21.8)
* Received curative surgery with one month
* Cancer stage I-III
* Age between 20 to 75
* Have an access to the internet at home

Exclusion Criteria:

* Diagnosed with severe psychological diseases or having a poor mental state preventing cooperate with research measures
* Not able to communicate verbally or with writing

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Functional Assessment of Cancer Therapy- Colorectal | Change from Baseline to 2, 4, and 6 months
  There are two subscales, 27 items of FACT-General and 9 items of Colorectal Cancer Subscale. Each item is rated on a 5-point Likert scale (0-4). The total score of the 36 items represents the score of the scale. The possible score for the scale ranges from 0 to 136. The higher values represent better quality of life.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline, 2, 4, and 6 months
  The Taiwan Version of International Physical Activity Questionnaire is used to measure a patient's physical activity. The scale has 7 items, asking patients the time they spent on walking, moderate, and vigorous physical activities during the past 7 days. The amounts of time spent on walking, moderate and vigorous physical activities are then multiplied by 3.3, 4.0, and 8.0 MET, respectively. The sum of the METs-min/wk for three types physically actives is the total score of the scale.
Cancer Behavior Inventory-Brief Version | Change from Baseline to 6 months
  There are 12 questions in total. It measures cancer patients 1) maintain independence and a positive attitude, 2) participate in medical care, (3) respond to and manage stress, and 4) Four aspects of self-efficacy, such as managing emotions. Each question is scored from 1 point "very unconfident" to 9 points "very confident". The total score of each question is the total score of the scale, and the possible range of scores Between 12 and 108 points, the higher the score, the higher the self-efficacy.
Supportive Care Needs Survey | Baseline, 2, 4, and 6 months
  34-item Supportive Care Needs Survey (SCNS-SF34) measures the supportive care needs of research subjects. This scale mainly to assess cancer patients' psychological (10 questions), health system and information (11 questions), body and daily life (5 questions), medical care and support ( 5 questions) and sex (3 questions) and other five aspects of support and care needs, each question is scored on a Lick-style scale ranging from 1 point "not necessary" to 5 points "very necessary", and the total score of each question is added. The total score in the table, the possible score ranges from 34 to 170 points, the higher the score, the higher the need for support and care.
M.D. Anderson Symptom Inventory | Baseline, 2, 4, and 6 months
  MDASI (M.D. Anderson Symptom Inventory) measures the symptom distress and consists of a 13-item symptom scale and a 6-item interference scale. The 13 symptoms were pain, fatigue, nausea, interrupted sleep, depression, shortness of breath, difficulty in remembering, loss of appetite, lethargy, dry mouth, sadness, vomiting, numbness/tingling. The interference scales for 6 questions are interference with walking, mobility, working ability (including housework), relationship with others, enjoying life, and mood. Each question is scored on a Lick-style scale ranging from 0 points "not at all" to 10 points "very bad". The average score of each question is the total score of the scale. The possible score ranges from 0 to 10 points. The higher the score, the more the symptom. The more serious the trouble, the average score of 1 to 4 means mild symptom distress, 5-6 means moderate symptom distress, and 7-10 means severe symptom distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (2):
- Taiwan (2):
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fridriksdottir N, Gunnarsdottir S, Zoega S, Ingadottir B, Hafsteinsdottir EJG. Effects of web-based interventions on cancer patients' symptoms: review of randomized trials. Support Care Cancer. 2018 Feb;26(2):337-351. doi: 10.1007/s00520-017-3882-6. Epub 2017 Sep 18. PMID 28921391
- [Background] Berry DL, Blonquist TM, Patel RA, Halpenny B, McReynolds J. Exposure to a patient-centered, Web-based intervention for managing cancer symptom and quality of life issues: impact on symptom distress. J Med Internet Res. 2015 Jun 3;17(6):e136. doi: 10.2196/jmir.4190. PMID 26041682